CLINICAL TRIAL: NCT04688307
Title: The Effect of Cigarette Smoking Reduction on Liver Function Tests and Metabolic Profile in Subjects With Non-alcoholic Steatohepatitis
Brief Title: Cigarette Smoking in Non-alcoholic Steatohepatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Raika Jamali, MD, Associate Professor of Medicine, Tehran University of Medical Sciences
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9411160001
Record Dates: First submitted 2019-11-01; First posted 2020-12-29 (Actual); Last update posted 2021-10-21 (Actual); Status verified 2021-10

CONDITIONS: Non-Alcoholic Fatty Liver Disease
Keywords: Steatohepatitis; Smoking; Aminotransferase
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Fatty Liver; Smoking | interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lifestyle modification and smoking reduction failure (Experimental): Obtaining ideal body weight by calorie restriction diet and programmed physical activity and the amount of cigarette smoking reduction is not more than 50% of the baseline
  Interventions: Behavioral: Motivational interviewing
- Lifestyle modification and smoking reduction (Experimental): Obtaining ideal body weight by calorie restriction diet and programmed physical activity and the amount of cigarette smoking reduction is 50% of the baseline or more
  Interventions: Behavioral: Motivational interviewing

INTERVENTIONS:
Behavioral: Motivational interviewing — Motivational interviewing for smoking reduction and adherence to diet and physical activity for obtaining ideal body weight

SUMMARY:
This non-randomized clinical trial was performed to clarify the effect of cigarette smoking reduction on liver function and some anthropocentric indices in smoker patients with non-alcoholic steatohepatitis.

DETAILED DESCRIPTION:
After excluding other causes of high aminotransferase level, participants with persistent elevated serum aminotransferase levels and evidence of fatty liver in ultrasonography were presumed to have non-alcoholic steatohepatitis. Those with NAFLD liver fat score greater than (-0.64) were enrolled. They were assigned to lifestyle modification alone or lifestyle modification plus smoking reduction groups.

Liver fat content, fasting serum glucose, alanine aminotransferase, aspartate aminotransferase, alkaline phosphatase, triglyceride, cholesterol, high and low-density lipoprotein, homeostasis model assessment-insulin resistance(HOMA-IR), and anthropometric measurements (body mass index and waist circumference) were checked at baseline and six months later.

ELIGIBILITY:
Inclusion Criteria:

Smokers with persistent elevated aminotransferase levels with the evidence of fatty liver in ultrasonography, who were referred to a gastroenterology clinic.

Exclusion Criteria:

* alcohol use (more than 20 gram per day in men and 10 gram per day in women per day),
* heart disease (ischemic or congestive),
* hepatic disease (viral hepatitis, autoimmune hepatitis, wilson disease, hemochromatosis, liver mass lesion),
* renal disease (serum creatinine concentration of > 1.5 mg/dl),
* any severe systemic co-morbidities, neoplasm,
* using any hepatotoxic medication during the past 3 months,
* pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Liver fat content percent change from baseline to 6 months | 6 months
  Liver fat content percent changes calculated by a formula

SECONDARY OUTCOMES:
Serum alanine aminotransferase level changes form baseline to 6 months | 6 months
  International unit per liter, Minimum value: 0, higher values show worse outcome

OTHER OUTCOMES:
Serum aspartate aminotransferase level changes form baseline to 6 months | 6 months
  International unit per liter, Minimum value: 0, higher values show worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Raika Jamali, MD, Principal Investigator — TUMS
Locations (2):
- Iran (2):
  - Gastroenterology clinic, Sina hospital., Tehran
  - Sina Hospital, TUMS, Tehran

IPD SHARING:
Plan to Share IPD: No